CLINICAL TRIAL: NCT06679855
Title: Milrinone for Prevention of Post-ligation Cardiac Syndrome Trial
Acronym: MIDAS
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: NICHD Neonatal Research Network (Network)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NICHD-NRN-0066
Record Dates: First submitted 2024-10-31; First posted 2024-11-08 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Post-ligation Cardiac Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): An iv infusion of placebo (0.9% saline) of equivalent volume will be administered. The infusion will be accompanied by an iv bolus of 10 mL/kg of 0.9% NaCl (administered over 60 minutes) to ensure blinding is maintained.
  Interventions: Drug: Placebo infusion
- Milrinone (Active Comparator): An intravenous (iv) infusion of milrinone will be administered at an initial dose of 0.33 mcg/kg/min and accompanied by an iv bolus of 10 mL/kg of 0.9% NaCl (administered over 60 minutes).
  Interventions: Drug: Milrinone infusion

INTERVENTIONS:
Drug: Milrinone infusion — An intravenous (iv) infusion of milrinone will be administered at an initial dose of 0.33 mcg/kg/min and accompanied by an iv bolus of 10 mL/kg of 0.9% NaCl (administered over 60 minutes).
  Arms: Milrinone
Drug: Placebo infusion — An iv infusion of placebo (0.9% saline) of equivalent volume will be administered. The infusion will be accompanied by an iv bolus of 10 mL/kg of 0.9% NaCl (administered over 60 minutes) to ensure blinding is maintained.
  Arms: Placebo

SUMMARY:
The goal of this Phase 3, randomized, masked clinical trial is to is to find out whether milrinone, when given to infants after PDA closure, will help the heart work better by supplying oxygen to the lungs and tissues.

The main questions it aims to answer are:

1. to determine if milrinone decreases the risk of death or PLCS within 7 days of the procedure, compared to standard treatment; and
2. to determine the effects of milrinone on two-year survival and neurodevelopmental outcome.

DETAILED DESCRIPTION:
Researchers will compare milrinone to a placebo saline solution to see if it helps the heart work better by supplying oxygen to the lungs and tissues.

After randomization the following will happen in both the control and treatment groups:

* Infant will start receiving either a low dose (0.33 μg/kg/min) of milrinone in the treatment group, OR saline solution in the control group through an intravenous (IV) line. The study drug will be started within 2 hours of the PDA closure procedure.
* For the first 2 to 4 hours, the study team will monitor very closely to see if there are any major side effects from the study drug.
* If the infant continues to have high blood pressure, which places an added stress on the heart, the dose will go up to 0.66 μg/kg/min. One more increase will be allowed to 0.75 μg/kg/min. The study drug will then stay at this dose. No more changes will happen to the dose. If there are side effects, then the study drug will be stopped and will not be started again.
* The study drug will be stopped after 24 hours if the infant only required the lowest drug and remains well. If the required higher doses of milrinone, it will take longer to wean them off the medication. Some infants may receive milrinone for 3-5 days. If the infant's heart starts to work better by using less oxygen from the breathing machine (ventilator), the study drug may be stopped before 3 days.
* Information will be collected from the infant's medical record including demographic information, gestational age, blood pressures, heart rates, respiratory rates, information about his or her breathing, medications, details of medical treatment for PDA, medical procedures including echocardiograms (ultrasound of the baby's heart), details of PDA closure (by surgery or transcatheter closure), head ultrasounds, and diagnoses. The investigators will also be collecting information from the maternal medical record including ultrasounds that may be relevant to the infant's course.
* Right after the study drug is stopped (which could be 5 days or less) the doctor may decide to give the infant the drug milrinone. This is a decision that will be made by the infant's doctor.
* After the infant goes home from the hospital, they will be scheduled for follow-up exams in the clinic. The follow-up visit will be done when the infant is about 2 years old. The visit will take about two hours to do. During the follow-up visit the investigators will test the infant's movement, behavior, and development. The investigators will also check the infant to make sure they do not have high blood pressure or any evidence of kidney disease.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age at birth ≤27 weeks (and 6 days) and postnatal age < 3 months at intervention
* Invasive or non-invasive positive pressure respiratory support (does not include low flow nasal cannula)
* Hemodynamically significant PDA with minimum transductal diameter ≥1.0 mm within 2 days of intervention
* Decision by clinical team to proceed with PDA closure via surgical ligation or percutaneous cardiac catheterization based on clinical and echocardiography features of hemodynamic significance.

Exclusion Criteria:

* Any major congenital malformation
* Congenital heart disease (except small (≤1mm) muscular ventricular septal defects, or small/moderate (<3mm) atrial septal defect)
* Acute renal failure defined by urine output < 0.5 mL/kg/hour OR rise of serum creatinine by 0.3 mg/dL within 48 hours OR rise of serum creatinine more than 40% above baseline serum creatinine within prior 72 hours.
* Systemic administration of vasodilator/inodilator agents
* Prior history of arrhythmia

Max Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 316 (Estimated)
Dates: Start 2025-06-13 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Post-ligation cardiac syndrome (PLCS) or death within 7 days of PDA closure | Onset within 48 hours but may last up to 7 days
  Composite outcome of post-ligation cardiac syndrome (PLCS) or death within 7 days of PDA closure. Onset within 48 hours but may last up to 7 days.

SECONDARY OUTCOMES:
Systemic hypotension | Onset within 48 hours but may last up to 7 days
  Either systolic blood pressure below the 3rd percentile for gestational age or mean blood pressure below the postmenstrual age equivalent
Systemic hypertension | Onset within 48 hours but may last up to 7 days
  Systolic blood pressure above the 97th percentile
Oxygenation failure | Onset within 48 hours but may last up to 7 days
  An absolute increase of at least 20% in the fraction of inspired oxygen or mean airway pressure compared with the one-hour post-intervention value that persists for a minimum of 1 hour and occurs within 72 hours of PDA closure
Ventilation failure | Within 72 hours of PDA closure
  Need for high frequency oscillatory ventilation when conventional ventilation strategies fail or a 20% rise in amplitude compared with the one-hour post-intervention value that persists for a minimum of 1 hour and occurs within 72 hours of PDA closure
Vasopressor score | Within 7 days of PDA closure
  Vasopressor score. Minimum score is zero. Higher score is worse, meaning need for higher level of support.
  VISmax will be calculated as follows: (VIS=dopamine dose [μg kg-1 min-1]+dobutamine [μg kg-1 min-1]+100×epinephrine dose [μg kg-1 min-1]+50×levosimendan dose [μg kg-1 min-1]+10×milrinone dose [μg kg-1 min-1]+10 000×vasopressin [units kg-1 min-1]+100×norepinephrine dose [μg kg-1 min-1]) using the maximum dosing rates of vasoactive and inotropic medications (μg kg-1 min-1 or IU kg-1 min-1)
Use of open-label milrinone or systemic vasodilator after cessation of study drug administration | After study drug cessation and within 7 days of PDA closure
  Number of participants using open-label milrinone or systemic vasodilator after cessation of study drug administration
Time to successful extubation | 36 weeks postmenstrual age
  Time to successful extubation, which is defined as extubation for at least 7 days
Post-intervention Moderate-severe bronchopulmonary dysplasia at 36 weeks' gestation | 36 weeks postmenstrual age
  Need for at least 2 liters of high flow nasal cannula at 36 weeks postmenstrual age
Post-intervention Chronic Pulmonary hypertension | 36 weeks postmenstrual age
  presence of septal flattening (or eccentricity index > 1.3, right ventricular systolic pressure greater than 40 mmHg, or exclusive right to left atrial level shunt on 36-week echocardiography assessment. The presence of a large atrial septal defect, pulmonary vein stenosis or left ventricular diastolic dysfunction will be recorded.
Post-intervention Periventricular Leukomalacia (PVL) | 36 weeks postmenstrual age
  Presence of cystic white matter changes on cranial ultrasound
Post-intervention Necrotizing Enterocolitis | 36 weeks postmenstrual age
  At least Bells stage IIb disease
Post-intervention Retinopathy of Prematurity (ROP) ≥ stage 3 (according to the international classification) | 36 weeks postmenstrual age
  Post-intervention Retinopathy of Prematurity (ROP) ≥ stage 3 (according to the international classification)
Weight or head circumference z-score change at 36 weeks | 36 weeks postmenstrual age
  Weight or head circumference z-score change at 36 weeks (decline by two z-scores will be considered growth failure)
Death between randomization and discharge from NICU | Randomization to 120 days' postnatal age, death, discharge, or transfer outside of the Study Center, whichever occurs first (an average of 112 days postnatal age)
  Death between randomization and discharge from NICU
Moderate-Severe neurodevelopmental impairment (NDI), using current NRN Follow-Up Study definition | 22 to 26 months
  Moderate-Severe neurodevelopmental impairment (NDI), using current NRN Follow-Up Study definition
Moderate-Severe neurodevelopmental impairment (NDI) or death | 22 to 26 months
  Moderate-Severe neurodevelopmental impairment (NDI) or death
Moderate or severe cerebral palsy | 22 to 26 months
  Moderate or severe cerebral palsy
Severe vision impairment | 22 to 26 months
  Severe vision impairment
Severe hearing impairment | 22 to 26 months
  Severe hearing impairment
Bayley-4 cognitive, language, motor scores | 22 to 26 months
  Bayley-4 cognitive, language, motor scores
Gross Motor Function level ≥II | 22 to 26 months
  Gross Motor Function level ≥II
CBCL Internalizing, Externalizing, and Total Problems aggregate T scores of >64 (clinical range) and 60-63 (borderline range). | 22 to 26 months
  CBCL Internalizing, Externalizing, and Total Problems aggregate T scores of >64 (clinical range) and 60-63 (borderline range).
Death before 22-26-month follow-up | 22 to 26 months
  Death before 22-26-month follow-up
Height, weight, or head circumference growth failure | 22 to 26 months
  Height, weight, or head circumference growth failure (decline by >2 z-scores since discharge)

CONTACTS AND LOCATIONS:
Locations (19):
- United States (19):
  - University of Alabama - Birmingham, Birmingham, Alabama
  - Children's Hospital of Orange County, Orange, California
  - Stanford University, Palo Alto, California
  - Sharp Mary Birch Hospital for Women & Newborns, San Diego, California
  - Emory University, Atlanta, Georgia
  - Northwestern Lurie Children's Hospital of Chicago, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - Boston Children's Hospital, Boston, Massachusetts
  - University of Mississippi Medical Center, Jackson, Mississippi
  - University of New Mexico, Albuquerque, New Mexico
  - Duke University, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - University of Oklahoma Health Sciences, Oklahoma City, Oklahoma
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Le Bonheur Children's Hospital, Memphis, Tennessee
  - University of Texas Southwestern, Dallas, Texas
  - University of Texas at Houston, Houston, Texas
  - University of Utah, Salt Lake City, Utah

REFERENCES:
- [Derived] McNamara PJ, Chock VY, Rahde-Bischoff A, Gabrio J, Johnson KJ, Harmon HM, Montoya-Williams D, Colaizy TT, Katheria AC, Ines F, Sorrells K, Battersby C, Levy PT, Rysavy MA, Bhombal S, Laughon MM, Carper B, Hintz SR, Das A, Bell EF. Evaluating the efficacy and safety of milrinone for prevention of post-patent ductus arteriosus closure syndrome (the MIDAS trial) in extremely preterm infants: a multicentre, double-masked, randomised, placebo-controlled trial. BMJ Open. 2025 Aug 26;15(8):e105018. doi: 10.1136/bmjopen-2025-105018. PMID 40858367